CLINICAL TRIAL: NCT01097863
Title: Clinical Validation of the New Print on Focus DAILIES Toric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-346-C-010
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- nelfilcon A, modified inversion indicator (Experimental): Nelfilcon A investigational contact lenses worn in both eyes on a daily wear, daily disposable basis for one week
  Interventions: Device: nelfilcon A contact lens, modified inversion indicator
- nelfilcon A, no inversion indicator (Experimental): Nelfilcon A investigational contact lenses worn in both eyes on a daily wear, daily disposable basis for one week
  Interventions: Device: nelfilcon A contact lens, no inversion indicator
- nelfilcon A, inversion indicator (Active Comparator): Nelfilcon A commercially marketed contact lenses worn in both eyes on a daily wear, daily disposable basis for one week.
  Interventions: Device: nelfilcon A contact lens, inversion indicator

INTERVENTIONS:
Device: nelfilcon A contact lens, modified inversion indicator — Investigational, nelfilcon A, toric, soft contact lens for daily disposable wear, with modified inversion indicator
  Arms: nelfilcon A, modified inversion indicator
Device: nelfilcon A contact lens, no inversion indicator — Investigational, nelfilcon A, toric, soft contact lens for daily disposable wear, with no inversion indicator
  Arms: nelfilcon A, no inversion indicator
Device: nelfilcon A contact lens, inversion indicator — Commercially marketed, nelfilcon A, toric, soft contact lens for daily disposable wear, with inversion indicator
  Other Names: Focus DAILIES Toric
  Arms: nelfilcon A, inversion indicator

SUMMARY:
The purpose of this study is to validate the improvements to the inversion indicator.

DETAILED DESCRIPTION:
This study was conducted in three countries under three separate protocols: P-346-C-009 sub 02 (UK), P-346-C-009 sub 03 (Germany), and P-346-C-010 (USA). The data reported represents pooled data from the three protocols.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age and sign written Informed Consent Document. If under legal age, parent or guardian must sign Informed Consent Document and subjects ages 12 through 17 must sign Informed Assent.
* Willing and able to wear study lenses in both eyes in the available parameters.
* Light-eyed subjects.
* Able to achieve 20/40 or better distance visual acuity (VA) in each eye at time of dispensing.
* Optimal or acceptable fit in each eye at time of dispensing.
* Willing to wear the study lenses at least 8 hours a day, 5 days a week.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks prior to enrollment for this trial.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in an ophthalmic clinical trial.
* Evidence of systemic or ocular abnormality, infection or disease which is likely to affect successful wear of contact lenses or use of their accessory solutions as determined by the investigator.
* Any use of medications for which contact lens wear could be contraindicated as determined by the investigator.
* RGP contact lens wearer.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This reporting group includes all enrolled and dispensed participants. Note: One subject was enrolled but not dispensed due to failing inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Nelfilcon A, Modified Inversion Indicator | Nelfilcon A, No Inversion Indicator | Nelfilcon A, Inversion Indicator
Started | 90 | 98 | 91
Completed | 89 | 98 | 89
Not Completed | 1 | 0 | 2
Not completed — Discomfort | 1 | 0 | 1
Not completed — Did not return for final visit | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nelfilcon A, Modified Inversion Indicator | Nelfilcon A, No Inversion Indicator | Nelfilcon A, Inversion Indicator | Total
Number analyzed (Participants) | 90 | 98 | 91 | 279
Age Continuous [Mean (Standard Deviation); unit: years] | 36.2 (10.6) | 33.3 (11.7) | 34.1 (10.8) | 34.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 69 | 69 | 190
  Male | 38 | 29 | 22 | 89

OUTCOME MEASURES:

1. Primary Outcome: Visibility of the Inversion Indicator on Lens When Lens Was on Participant's Finger, for Example, During Lens Insertion.
Description: As assessed by the participant retrospectively after one week of wear and recorded on a questionnaire as a yes or no response to the question, "Did you notice an OK mark on the study lens while it was on your finger, for example, during lens insertion?" The positive "yes" responses are reported.
Time Frame: 1 week
Population: Analysis conducted per protocol, with exclusions due to protocol deviations as determined by masked review (9), and unavailable data due to discontinuations (3).
Measure: Number; unit: participants
Arm/Group | Nelfilcon A, Modified Inversion Indicator | Nelfilcon A, No Inversion Indicator | Nelfilcon A, Inversion Indicator
Number analyzed (Participants) | 86 | 97 | 84
participants | 77 | 15 | 84

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the trial: 78 days
Description: This reporting group includes all enrolled and exposed participants: 280
Arm/Group | Nelfilcon A, Modified Inversion Indicator | Nelfilcon A, No Inversion Indicator | Nelfilcon A, Inversion Indicator
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/98 | 0/92
Other Adverse Events (participants affected / at risk) | 6/90 | 13/98 | 13/92
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelfilcon A, Modified Inversion Indicator (N=90) | Nelfilcon A, No Inversion Indicator (N=98) | Nelfilcon A, Inversion Indicator (N=92)
Other contact lens symptoms not requiring treatment (Eye disorders) | 6 (6) | 13 (13) | 13 (13) — Participants reported on a questionnaire the nature, frequency and severity of any/all lens-related symptoms experienced with lens wear. Any frequency and/or severity significantly higher with study lenses than with habitual was an adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussion, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.